CLINICAL TRIAL: NCT00774839
Title: A Study of Economic Circumstances, Service Utilization, and Service Needs Among Older Colon Cancer Patients
Brief Title: Study of Economic Circumstances, Service Utilization, and Service Needs Among Older Colon Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); State University of New York - Downstate Medical Center (Other); Ralph Lauren Center for Cancer Care and Prevention (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 08-124
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer
Keywords: Newly Diagnosed; Colon; Stage II; Stage III
MeSH Terms: conditions — Colonic Neoplasms | interventions — Demography; Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Newly diagnosed stage II-III colon cancer 65 years or older: Medicare-eligible (≥ or = to 65 years) patients diagnosed with stage II - III colon cancer, are at least 4 months into chemotherapy and up to 7 months post-chemotherapy.
  Interventions: Behavioral: Patient Interview

INTERVENTIONS:
Behavioral: Patient Interview — The patient will participate in a semistructured interview conducted by a trained staff member and designed to last approximately 45 minutes. All interviews will take place at least 4 months into or up to 7 months after the end of the treatment, if possible and will be scheduled to occur at the time of the chemotherapy infusion, or at another time at the care facility when it is convenient for the patient. If the patient is not scheduled or chooses not to be at the care facility within a time frame that fits the study parameters, the patient may opt to be interviewed at another location, including the patient's home.
  Other Names: The interview includes five major topic areas: 1) Demographics and Health; 2) Expenses;; 3) Utilization of Supports and Services; 4) Impact on Financial and Social Well-Being;; and 5) Unmet Resources/Service Needs.

SUMMARY:
The purpose of this study is to learn more about the social and financial impact of colon cancer for older patients. We want to know how cancer has affected the patient financially and socially, and to know if the patient has resource needs that have gone unmet. By doing this study, we hope to learn about resources that can reduce the financial burden from cancer.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Newly diagnosed stage II-III colon cancer
* Receiving chemotherapy and at least 4-6 months into chemotherapy treatment, or have received chemotherapy and no more than 7 months post-treatment
* Sufficient cognitive capacity as determined by investigator or consenting professional
* Able to speak English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* N/A

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will be recruiting from eight sites of care that serve different populations, which will allow us to sample Medicare-eligible individuals with a range of income, insurance coverage and socio-demographic characteristics. These sites are: Memorial Sloan-Kettering Cancer Center (MSKCC); four MSKCC Network locations (Commack, Phelps,Mercy, and Basking Ridge); SUNY Downstate Medical Center;Ralph Lauren Cancer Center and Albert Einstein College of Medicine/Montefiore Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Self-reported expenses associated with colon cancer treatment and living with this illness. | conclusion of study

SECONDARY OUTCOMES:
The perceived impact of cancer on patients' overall financial and social well-being. | conclusion of study
The awareness of cancer support organizations and their utilization of informal and formal supports during treatment. | conclusion of study
The patients' unmet resource and service needs during treatment. | conclusion of study
Identify the medical, social and economic risk factors that are most closely associated with perceived adverse impact on financial and social well-being and unmet resource and service needs. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Elena Elkin, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org